CLINICAL TRIAL: NCT07142408
Title: The Effect of Pre-Operative Bacterial Decolonization on Post-Operative Infection Rate for Lower Extremity Wounds Healing by Second Intention
Brief Title: The Effect of Bacterial Decolonization Before Skin Cancer Surgery on Infection Rate of Lower Extremity Wounds Left Open to Heal
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: University of California, Davis (Other); Washington University School of Medicine (Other); Baylor College of Medicine (Other); Princeton Healthcare System (Other); The Cleveland Clinic (Other); University of Georgia (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cooper IRB Number 21-119
Record Dates: First submitted 2025-07-29; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Surgical Wound Infection
Keywords: Lower Extremity Wound; Skin Cancer Surgery; Infection Rate; Prophylactic Topical Antibiotics; Chlorhexidine; Mupirocin; Wound Healing; Secondary Intention; Infection Prevention
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; Mupirocin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): This group will be prophylactically treated with topical antibiotics every day for 5 days prior to surgery. Participants will shower with Hibiclens antiseptic skin cleanser once daily and apply mupirocin ointment to the nares twice daily, in the morning and evening.
  Interventions: Drug: Chlorhexidine gluconate (4%); Drug: Mupirocin 2% Ointment
- Control Group (No Intervention): This group will NOT be prophylactically treated with Hibiclens antiseptic skin cleanser and mupirocin ointment prior to surgery.

INTERVENTIONS:
Drug: Chlorhexidine gluconate (4%) — Chlorhexidine 4% solution will be applied from the neck down (avoiding the face, penis, and vagina), allowed to sit on the skin for one minute, then rinsed off in the shower every day for 5 days prior to surgery.
  Other Names: Hibiclens
  Arms: Treatment Group
Drug: Mupirocin 2% Ointment — Mupirocin 2% ointment will be applied to the inside of the nostrils twice daily, in the morning and evening, for 5 days prior to surgery. A small amount of the ointment will be placed on the tip of a cotton swab to facilitate application to each nostril.
  Arms: Treatment Group

SUMMARY:
The goal of this clinical trial is to learn if reducing bacterial load on the skin and nostrils with topical antibacterial soap and ointment, respectively, reduces rate of infection in surgical sites on lower leg wounds left open to heal in adults undergoing skin cancer surgery.

The main question it aims to answer is:

Does Hibiclens antibacterial skin cleanser and mupirocin antibacterial ointment applied to nostrils prior to surgery lower the number of times participants develop an infection in their open wound on the lower leg?

Researchers will compare the treatment group to the standard of care, which involves no treatment prior to surgery, to see if topical antibiotics applied prior to surgery affect infection rates between the two groups.

Participants randomized to the treatment group will:

Shower with Hibiclens once daily for 5 days prior to the day of surgery and apply mupirocin to the nostrils twice daily for 5 days prior to the day of surgery. They will then send pictures of their surgical site to monitor for signs of infection at 2-week and 4-week post-operation.

Participants randomized to the control group (standard of care) will:

NOT apply the topical antibacterials prior to the day of surgery. They will then send pictures of their surgical site to monitor for signs of infection at 2-week intervals for 1 month after surgery.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if reducing bacterial load on the skin and nostrils with topical antibacterial soap and ointment, respectively, reduces rate of infection in surgical sites on lower leg wounds left open to heal in adults undergoing skin cancer surgery.

The main question it aims to answer is:

Does Hibiclens antibacterial skin cleanser and mupirocin ointment applied to nostrils prior to surgery lower the number of times participants develop an infection in their open wound on the lower leg?

Researchers will compare the treatment group to the standard of care, which involves no treatment prior to surgery, to see if topical antibiotics applied prior to surgery affect infection rates between the two groups.

Participants randomized to the treatment group will:

1. Shower with Hibiclens (Chlorhexidine Gluconate Solution 4% w/v) once daily for 5 days prior to the day of surgery
2. Apply 2% mupirocin ointment to the nostrils twice daily for 5 days prior to the day of surgery
3. Come into the office for their skin cancer surgery. They will be provided with standard wound care instructions, which entails daily gentle cleansing with soap/water, pat dry, then apply Vaseline, nonadherent gauze, and paper tape.
4. Send pictures of their surgical site at 2-week and 4-week post-operation, which will be monitored for signs of infection by the study physicians.
5. If there's a concern for infection, they will come into the office to swab the wound site to determine the cause of infection. If there's no concern for infection, they will not need to return to the office.

Participants randomized to the control group (standard of care) will:

1. NOT apply the topical antibacterials prior to the day of surgery
2. Come into the office for their skin cancer surgery. They will be provided with standard wound care instructions, which entails daily gentle cleansing with soap/water, pat dry, then apply Vaseline, nonadherent gauze, and paper tape.
3. Send pictures of their surgical site at 2-week and 4-week post-operation, which will be monitored for signs of infection by the study physicians.
4. If there's a concern for infection, they will come into the office to swab the wound site to determine the cause of infection. If there's no concern for infection, they will not need to return to the office.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Scheduled to undergo surgical treatment for skin cancer on the lower extremities and have no other surgeries scheduled in the coming weeks after the procedure
* Will have a surgical wound that will be left open to heal by secondary intention

Exclusion Criteria:

* Age under 18 years old
* Have a known allergy to chlorhexidine or mupirocin
* Have a history of Staphylococcus aureus infection
* Have a history of heart valve or joint replacement surgery requiring pre-operative antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Surgical Site Wound Infection | From date of surgery to 1-month post-operation
  Signs of infection, including erythema, edema, drainage, and delayed healing, will be visually determined by study physicians with photographs of the surgical site collected from study participants. All patients will be followed up with a phone call at 1 month to monitor for any adverse events and additional signs of infection including pain, tenderness, warmth, and foul odor at the surgical site.

SECONDARY OUTCOMES:
Type of Pathogens Present in Surgical Site | From date of surgery to 1-month post-operation
  Study participants with signs of infection, as determined by the study physicians from photos of the wound, will return to the office for a wound culture to determine the type of pathogen causing the infection.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Dermatologic Surgery at Cooper University Health Care, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided whether or not individual participant data (IPD) will be shared, however, if we do, only IPD used in the results publication will be included.

REFERENCES:
- [Background] Smith H, Borchard K, Cherian P, Tai Y, Vinciullo C. Randomized Controlled Trial of Preoperative Topical Decolonization to Reduce Surgical Site Infection for Staphylococcus aureus Nasal Swab-Negative Mohs Micrographic Surgery Patients. Dermatol Surg. 2019 Feb;45(2):229-233. doi: 10.1097/DSS.0000000000001662. PMID 30204741
- [Background] Cherian P, Gunson T, Borchard K, Tai Y, Smith H, Vinciullo C. Oral antibiotics versus topical decolonization to prevent surgical site infection after Mohs micrographic surgery--a randomized, controlled trial. Dermatol Surg. 2013 Oct;39(10):1486-93. doi: 10.1111/dsu.12318. PMID 24090258
- [Background] Molina GE, Yu SH, Neel VA. Observations Regarding Infection Risk in Lower-Extremity Wound Healing by Second Intention. Dermatol Surg. 2020 Oct;46(10):1342-1344. doi: 10.1097/DSS.0000000000002094. No abstract available. PMID 31415257
- [Background] Dixon AJ, Dixon MP, Askew DA, Wilkinson D. Prospective study of wound infections in dermatologic surgery in the absence of prophylactic antibiotics. Dermatol Surg. 2006 Jun;32(6):819-26; discussion 826-7. doi: 10.1111/j.1524-4725.2006.32167.x. PMID 16792648
- [Background] Liu X, Sprengers M, Nelemans PJ, Mosterd K, Kelleners-Smeets NWJ. Risk Factors for Surgical Site Infections in Dermatological Surgery. Acta Derm Venereol. 2018 Feb 7;98(2):246-250. doi: 10.2340/00015555-2844. PMID 29136259
- [Background] Schimmel J, Belcher M, Vieira C, Lawrence N, Decker A. Incidence of Surgical Site Infections in Second Intention Healing After Dermatologic Surgery. Dermatol Surg. 2020 Dec;46(12):1492-1497. doi: 10.1097/DSS.0000000000002409. PMID 32483093

DOCUMENTS (1):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT07142408/Prot_000.pdf